CLINICAL TRIAL: NCT04047069
Title: The Effect of Person-Centered Occupational Therapy Intervention on Occupational Performance and Quality of Life in Hemodialysis Patients
Brief Title: The Effect of Occupational Therapy Intervention in Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/257
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Quality of Life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Awareness Training
  Interventions: Behavioral: Awareness Training
- Intervention group (Experimental): * Awareness Training
  * Person-Centered Occupational Therapy Intervention
  Interventions: Behavioral: Awareness Training and Person-Centered Occupational Therapy Intervention

INTERVENTIONS:
Behavioral: Awareness Training and Person-Centered Occupational Therapy Intervention — Exp. identifying the activities the person wants to do, suggestions to facilitate the activity, arranging the activity according to the needs of the person, arranging the environment so that the environment can be a facilitating factor in the activities the person wants to do.
  Arms: Intervention group
Behavioral: Awareness Training — Exp.
  * General information about HD
  * Approaches to Coping with HD Symptoms
  * Self care skills (eg hygiene)
  Arms: Control

SUMMARY:
The aim of this study is to investigate the effect of person-centre occupational therapy intervention on activity performance and quality of life in hemodialysis patients. The results of the study will guide the intervention programs for prevention, coping and improving the quality of life of HD patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as chronic renal failure.
* between 18-65 years
* undergoing HD treatment for at least 1 year

Exclusion Criteria:

* Beck Depression Scale score of 17 or higher

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-12 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life (with a quality of life scale specific to renal patients). | 1st day of study
  The KidneyDisease Quality of Life (KDQOL-36) consists of the SF-12, which measures physical and mental functioning, Burden of Kidney Disease subscale, Symptoms and Problems subscale, and Effects of Kidney Disease on Daily Life subscale. The scores of theKDQOL-36 questionnaire are transformed into 0 to 100, with higherscores indicating better quality of life.combines the generic SF-36 Health Survey instrument and disease-specific components for assessing the health-related quality of life of

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Trakya University
Locations (1):
- Özgü İnal, Edirne, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No